CLINICAL TRIAL: NCT05794464
Title: Secretoneurin as a Biomarker of Atrial Fibrillation rEcurrence After Catheter Ablation/Electrical Cardioversion
Brief Title: The SAFE Prospective Registry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FNO-IKK-SAFE
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation, Paroxysmal or Persistent
Keywords: atrial fibrillation; secretoneurin; catheter ablation; electrical cardio version
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled in one group.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catheter ablation and/or electrical cardioversion (Experimental): Study subjects indicated for catheter ablation and/or electrical cardioversion will be enrolled in this study arm.
  Interventions: Procedure: Catheter ablation and/or electrical cardioversion

INTERVENTIONS:
Procedure: Catheter ablation and/or electrical cardioversion — Catheter ablation and/or electrical cardio version are procedures intended to treat atrial fibrillation.

SUMMARY:
Secretoneurin (SN) is a neuropeptide from the chromogranin family that influences intracellular calcium handling. SN suppresses calcium leakage from the sarcoplasmic reticulum through the ryanodine receptor. SN is a novel biomarker that has shown the potential to predict adverse arrhythmic events.

DETAILED DESCRIPTION:
The aim of the study is to sample SN before and after catheter ablation (CA) for atrial fibrillation (Afib) to predict the recurrence after CA. Also, the uric acid/albumin ratio will be assessed as a marker of Afib recurrence. Since the uric acid/albumin ratio has been shown to be predictive of Afib in patients with myocardial infarction moreover incidence of atrial fibrillation is higher in patients with gout. As a side branch marker for silent brain injury, neuron-specific enolase (NSE) and protein S100B will be evaluated. NSE showed in small trials a significant increase after catheter ablation, as well as S100B. The prognostic power is not clear yet. From the systematic review, the most powerful predictors seem to be N-terminal (NT)-prohormone B-type natriuretic peptide (NT-Pro-BNP/BNP), high-sensitivity C-reactive protein (hs-CRP), interleukin-6 (IL-6) and Carboxy-terminal telopeptide of collagen type I. Biomarkers are divided into 3 main types: congestion, inflammation, and renal function.

Patients will be enrolled before catheter ablation/electrical cardioversion for Afib after signing IS, and the blood sampling will be performed the day before and the day after catheter ablation. In the electric cardioversion arm, the blood sampling will be performed before electrical cardioversion and 2h after the cardioversion before discharge.

Patients will be followed for recurrency - all patients will have a 24-hour ECG Holter and External loop recorder (MDT) for two weeks after the three months of the blanking period. Clinical outpatient control will ensue in the 4th, eighth,12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation (Afib); (paroxysmal, persistent)
* Patients indicated for catheter ablation and/or electrical cardioversion
* Signed informed consent

Exclusion Criteria:

* Longstanding or permanent atrial fibrillation
* Severe mitral regurgitation
* Heart failure with a permanently reduced ejection fraction
* Cerebral ischaemic stroke in < 3 months
* Severe kidney injury
* Severe renal insufficiency
* Hepatic insufficiency limiting biomarker sampling
* Myocardial infarction < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence based on secretoneurin levels | 24 months
  Atrial fibrillation recurrence based on secretoneurin levels will be assessed

SECONDARY OUTCOMES:
Brain injury detection | 24 months
  Brain injury will be detected using serum protein S100B and neuron specific enolase.

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Plášek, MD,PhD,FESC, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Anderson ME. Will secretoneurin be the next big thing? J Am Coll Cardiol. 2015 Feb 3;65(4):352-354. doi: 10.1016/j.jacc.2014.11.028. No abstract available. PMID 25634833
- [Background] Ottesen AH, Louch WE, Carlson CR, Landsverk OJB, Kurola J, Johansen RF, Moe MK, Aronsen JM, Hoiseth AD, Jarstadmarken H, Nygard S, Bjoras M, Sjaastad I, Pettila V, Stridsberg M, Omland T, Christensen G, Rosjo H. Secretoneurin is a novel prognostic cardiovascular biomarker associated with cardiomyocyte calcium handling. J Am Coll Cardiol. 2015 Feb 3;65(4):339-351. doi: 10.1016/j.jacc.2014.10.065. PMID 25634832
- [Background] Selcuk M, Cinar T, Saylik F, Akbulut T, Asal S, Cicek V, Hayiroglu MI, Tanboga IH. Predictive value of uric acid/albumin ratio for the prediction of new-onset atrial fibrillation in patients with ST-Elevation myocardial infarction. Rev Invest Clin. 2022 May 2;74(3):156-164. doi: 10.24875/RIC.22000072. PMID 35797660
- [Background] Zhong X, Jiao H, Zhao D, Teng J. Serum Uric Acid Levels in Relation to Atrial Fibrillation: A Case-Control Study. Med Sci Monit. 2022 Feb 27;28:e934007. doi: 10.12659/MSM.934007. PMID 35220390
- [Background] Kuo YJ, Tsai TH, Chang HP, Chua S, Chung SY, Yang CH, Lin CJ, Wu CJ, Hang CL. The risk of atrial fibrillation in patients with gout: a nationwide population-based study. Sci Rep. 2016 Sep 7;6:32220. doi: 10.1038/srep32220. PMID 27599578
- [Background] Acibuca A, Vurgun VK, Gerede DM, Altin AT, Gul IS, Candemir B, Isikay Togay C, Kilickap M, Akyurek O. Serum neuron-specific enolase, a marker of neuronal injury, increases after catheter ablation of atrial fibrillation. J Int Med Res. 2018 Nov;46(11):4518-4526. doi: 10.1177/0300060518767768. Epub 2018 Sep 5. PMID 30185093
- [Background] Boyalla V, Harling L, Snell A, Kralj-Hans I, Barradas-Pires A, Haldar S, Khan HR, Cleland JGF, Athanasiou T, Harding SE, Wong T. Biomarkers as predictors of recurrence of atrial fibrillation post ablation: an updated and expanded systematic review and meta-analysis. Clin Res Cardiol. 2022 Jun;111(6):680-691. doi: 10.1007/s00392-021-01978-w. Epub 2022 Jan 9. PMID 34999932
- [Derived] Plasek J, Vrtal J, Chobolova N, Svagera Z, Drienikova D, Pudich J, Rachela M, Stejskal D, Dodulik J, Vaclavik J. Secretoneurin plasma levels are decreased after catheter ablation for atrial fibrillation-patients with AF produce lower SN levels than healthy individuals: the SAFE registry. Front Cardiovasc Med. 2025 Oct 16;12:1664855. doi: 10.3389/fcvm.2025.1664855. eCollection 2025. PMID 41179559